CLINICAL TRIAL: NCT04674761
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of Odevixibat (A4250) in Patients With Alagille Syndrome (ASSERT)
Brief Title: Efficacy and Safety of Odevixibat in Patients With Alagille Syndrome
Acronym: ASSERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4250-012
Record Dates: First submitted 2020-12-10; First posted 2020-12-19 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Alagille Syndrome
Keywords: ALGS; Alagille syndrome
MeSH Terms: conditions — Alagille Syndrome | interventions — odevixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odevixibat (A4250) (Experimental): Capsules for oral administration once daily for 24 weeks.
  Interventions: Drug: Odevixibat
- Placebo (Placebo Comparator): Capsules for oral administration (to match active) once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Odevixibat — Odevixibat is a small molecule and selective inhibitor of IBAT.
  Other Names: A4250
  Arms: Odevixibat (A4250)
Drug: Placebo — Placebo identical in appearance to experimental drug (odevixibat).
  Arms: Placebo

SUMMARY:
Double-blind, randomized, placebo-controlled, Phase 3 study to investigate the efficacy and safety of odevixibat compared to placebo in Patients with Alagille Syndrome.

DETAILED DESCRIPTION:
Approximately 35 sites will be initiated for this study in North America, Europe, Middle East, and Asia Pacific.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetically confirmed diagnosis of Alagille syndrome
* History of significant pruritus as measured by the Albireo Observer or Patient Reported Outcome instrument
* Elevated serum bile acid level

Key Exclusion Criteria:

* History or ongoing presence of other types of liver disease (eg. biliary atresia, progressive familial intrahepatic cholestasis, hepatocellular carcinoma)
* History of liver transplant, or a liver transplant is planned within 6 months of randomization
* ALT >10× upper limit of normal (ULN) at screening
* Total bilirubin >15 × ULN at screening
* Patient suffers from uncontrolled, recalcitrant pruritic condition other than Alagille syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (9):
  - University of California - San Francisco, San Francisco, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Childrens Hospital at Montefiore Albert Einstein School of Medicine, The Bronx, New York
  - Oregon Health Science University School of Medicine, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Cliniques Universitaires Saint-Luc Bruxelles, Brussels, Belgium
- CHU Sainte-Justine, Montreal, Quebec, Canada
- France (4):
  - Hôpital Femme Mère Enfant de Lyon, Bron
  - Antenne pédiatrique du CIC - Hopital Jeanne De Flandre, Lille
  - APHM, Marseille
  - Hopital Necker Enfants Malades, Paris
- Germany (3):
  - Charité-Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinik für Kinder-und Jugendmedizin Tübingen, Tübingen
- Israel (2):
  - Sharie Zedek, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (4):
  - ASST Papa Giovanni XXIII, Bergamo
  - AOU Meyer, Florence
  - Azienda Ospedale Università Padova, Padua
  - Bambino Gesù Children's Hospital, Rome
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - University Medical Centre Utrecht, WKZ, Utrecht
- Starship Child Health, Auckland, New Zealand
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- Turkey (Türkiye) (2):
  - Hacettepe Üniversitesi İhsan Doğramacı Çocuk Hastanesi, Ankara
  - Istanbul University Medical Faculty Hospital, Fatih
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Ovchinsky N, Aumar M, Baker A, Baumann U, Bufler P, Cananzi M, Czubkowski P, Durmaz O, Fischer R, Indolfi G, Karnsakul WW, Lacaille F, Lee WS, Maggiore G, Rosenthal P, Ruiz M, Sokal E, Sturm E, van der Woerd W, Verkade HJ, Wehrman A, Clemson C, Yu Q, Ni Q, Ruvido J, Manganaro S, Mattsson JP. Efficacy and safety of odevixibat in patients with Alagille syndrome (ASSERT): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2024 Jul;9(7):632-645. doi: 10.1016/S2468-1253(24)00074-8. Epub 2024 Apr 23. PMID 38670135

RESULTS

PARTICIPANT FLOW:
Groups:
- Odevixibat (A4250): Capsules for oral administration once daily for 24 weeks (120 μg/kg/day).
  Odevixibat: Odevixibat is a small molecule and selective inhibitor of IBAT.
Period: Overall Study
Arm/Group | Odevixibat (A4250) | Placebo
Started | 35 | 17
Completed | 35 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Odevixibat (A4250) | Placebo | Total
Number analyzed (Participants) | 35 | 17 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 17 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.73 (3.780) | 5.40 (4.411) | 6.29 (4.003)
Age, Customized [Count of Participants; unit: Participants]
  < 10 years | 29 | 13 | 42
  > = 10 years and < 18 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 21 | 6 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 13 | 43
  Black or African American | 2 | 2 | 4
  Asian | 2 | 1 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11
  United Kingdom | 1 | 0 | 1
  Malaysia | 2 | 1 | 3
  Netherlands | 3 | 3 | 6
  Turkey | 1 | 0 | 1
  Belgium | 1 | 1 | 2
  Poland | 7 | 3 | 10
  Italy | 4 | 2 | 6
  France | 3 | 1 | 4
  Germany | 6 | 2 | 8
Genetic Mutation [Count of Participants; unit: Participants]
  JAG1 | 32 | 16 | 48
  NOTCH2 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Scratching Score
Description: Change from baseline in average AM (measured after waking up) and PM (measured before bedtime) scratching score to Month 6 as measured by the Albireo Observer-Reported Outcome (ObsRO) Instrument. The ObsRO instrument was used to assess severity of observed scratching twice a day (AM and PM) with scores from 0 to 4 where 0 is no scratching and 4 is worst possible scratching.
Time Frame: Change from baseline for each four-week average pruritis score to Month 6 (Weeks 21 to 24), in which baseline was calculated based on the 14 days before the start of treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Odevixibat (A4250) | Placebo
Number analyzed (Participants) | 35 | 17
score on a scale | -1.69 (0.174) | -0.8 (0.233)
Statistical Analysis 1: Comparison: Odevixibat (A4250) vs Placebo; The analysis is based on a mixed model for repeated measures (MMRM) using a restricted maximum likelihood (REML) with baseline score as a covariate, and baseline age stratification, baseline direct bilirubin, treatment group, time (in months), and treatment-by-time interaction as fixed effects. One-sided p-value was reported; Test type: Superiority; p = 0.0012, Mixed Models Analysis; LS mean difference = -0.88, 95% CI 2-sided [-1.44 to -0.33], Standard Error of Mean 0.277

2. Secondary Outcome: Serum Bile Acid Levels
Description: Change in serum bile acid levels (μmol/L) from baseline to average of week 20 and 24
Time Frame: Change from baseline to average of week 20 and 24, where baseline was calculated by averaging the last two values preceding start of treatment, and average of Week 20 and Week 24 was defined as the average of Week 20 and Week 24 values.
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Odevixibat (A4250) | Placebo
Number analyzed (Participants) | 35 | 17
μmol/L | -90.35 (21.336) | 22.39 (28.463)
Statistical Analysis 1: Comparison: Odevixibat (A4250) vs Placebo; The analysis is based on a mixed model for repeated measures (MMRM) using a restricted maximum likelihood (REML) with baseline serum bile acid (sBA) concentration data as a covariate, and baseline age stratification, treatment group, visits (Weeks 4, 8, 12, 16, 20, 24), and treatment-by-visit interaction as fixed effects. The comparison of treatment difference in change from baseline to the average of Week 20 and Week 24 is estimated and tested using contrast. One-sided p-value was reported; Test type: Superiority; p = 0.0006, Mixed Models Analysis; LS mean difference = -112.74, 95% CI 2-sided [-178.78 to -46.69], Standard Error of Mean 32.864

ADVERSE EVENTS:
Time Frame: The safety reporting period for adverse events is from the first dose of study drug through the last planned study visit or 28 calendar days after the last dose of the study drug, whichever occurs later, up to 203 days.
Arm/Group | Odevixibat (A4250) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/17
Serious Adverse Events (participants affected / at risk) | 5/35 | 2/17
Other Adverse Events (participants affected / at risk) | 26/35 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odevixibat (A4250) (N=35) | Placebo (N=17)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odevixibat (A4250) (N=35) | Placebo (N=17)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 4 (7)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)
Conjunctivitis (Infections and infestations) | 2 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Vitamin A decreased (Investigations) | 1 (1) | 0 (0)
Vitamin E decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Albireo will retain the ownership of all data. All proposed publications based on this study must be subject to the sponsor's approval requirements.

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT04674761/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04674761/SAP_001.pdf